CLINICAL TRIAL: NCT00036426
Title: Phase II Study of FavId (Tumor-Specific Idiotype-KLH) and Soluble GM-CSF Immunotherapy in Patients With Stable or Progressive Grade 1 and 2 Follicular B-Cell Lymphomas
Brief Title: Idiotype Vaccine for Low-Grade Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Favrille (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FavId-01; NCT00014157 (obsolete NCT alias)
Record Dates: First submitted 2002-05-09; First posted 2002-05-10 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Lymphoma, Low-Grade
Keywords: lymphoma; vaccine; idiotype; KLH; GM-CSF
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Immunotherapy, Active

INTERVENTIONS:
Biological: FavId (Id-KLH) active immunotherapy

SUMMARY:
The purpose of this study was to determine if an idiotype vaccine, made from a patient's lymphoma that has returned after chemotherapy and/or rituximab, would be able to shrink their tumor.

DETAILED DESCRIPTION:
The purpose of this study was to assess the ability of active immunotherapy to induce tumor regressions in relapsed low-grade lymphoma. B-cell malignancies express a unique antigen, the immunoglobulin idiotype (Id), on their surface. Each B-cell harbors a unique genetic sequence used in the production of immunoglobulin idiotype. B-cell lymphomas arise from the clonal expansion of a single B-cell and all tumor cells express that unique Id protein. No normal B-cells possess that Id on their cell surface. Hence, Id protein should serve as an ideal target for individualized active immune therapy of NHL. Many of the antigens expressed by tumors (including Id) are only weak immunogens. To augment the immune response against Id, the Id protein must be chemically coupled to a strongly immunogenic protein. Keyhole limpet hemocyanin (KLH) is a commonly used protein carrier capable of augmenting the body's immune reaction against Id protein. While initial studies reported a predominately humoral (antibody) response, cellular immunity (T-cells) also plays a critical role in anti-tumor immunity. GM-CSF is a hematopoietic growth factor that stimulates T-cell proliferation.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age
* Histologically confirmed grade 1 or 2 follicular B-cell lymphoma (WHO classification)
* Patients that have responded with at least stable disease to their most recent chemo- or anti-CD20 antibody (Rituxan®, Zevalin, Bexxar) therapy for a minimum of 90 days and who currently have relapsed or who continue to have stable disease.
* Tumor accessible for biopsy or previously existing biopsy material
* At least 1 additional bidimensional lesion measuring at least 2 cm in each dimension
* Performance status (ECOG) of 0, 1 or 2
* Absolute Granulocyte count ? 1,000/mm3
* Total Bilirubin < 2 mg/dL
* AST and ALT < 2x Upper Limit of Normal
* Creatinine < 1.5 mg/dL

Exclusion Criteria

* Patients who have had more than 3 prior chemotherapy or anti-CD20 regimens
* Prior fludarabine
* Prior tumor-specific idiotype immunotherapy
* Patients whose disease has progressed within the first 90 days of their last chemotherapy or anti-CD20 treatment
* Concurrent immunosuppressive therapy (high-dose steroids; etc)
* Prior splenectomy
* Surgery, cancer radiotherapy, steroid therapy, immunotherapy or chemotherapy within 90 days prior to first scheduled vaccination
* Known history of CNS lymphoma or meningeal lymphomatosis
* HIV positive
* Serious non-malignant disease (e.g., psychiatric disorders, congestive heart failure, or active uncontrolled bacterial, viral, or fungal infections), or other conditions which, in the opinion of the investigator would compromise protocol objectives
* Prior malignancy (excluding nonmelanoma carcinomas of the skin and in situ cervical carcinomas) unless in remission for > 2 years
* Treatment with an investigational drug within 30 days prior to study entry
* Pregnant or nursing women NOTE: Women of childbearing potential should be advised to avoid becoming pregnant while receiving treatment with FavId.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2001-03

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Scripps Stevens Cancer Center, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - Oncology Associates of San Diego, San Diego, California
  - Medical Group of North County, Vista, California
  - University of Florida, Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - New York Hospital - Cornell Medical Center, New York, New York
  - New York Medical College - Our Lady of Mercy Medical Center, Comprehensive Cancer Center, The Bronx, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania